CLINICAL TRIAL: NCT03776877
Title: Evaluation of Clinical and Imaging Criteria, and Plasma Biomarkers of Patients Receiving an Endovascular Treatment for an Acute Ischemic Stroke
Brief Title: Endovascular Treatment in Ischemic Stroke Follow-up Evaluation
Acronym: ETIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2017024F
Record Dates: First submitted 2018-09-10; First posted 2018-12-17 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arterial Ischemic Stroke (AIS): All patients (prospective and retrospective) included will have to present an Arterial Ischemic Stroke (AIS) from a large cerebral vessel occlusion.
  The participation in the study will consist in:
  * Plasmatic collection at the time of AIS, for study of plasma biomarkers
  * Additional standardized blinded clinical evaluation at three months after the thrombectomy realized during a phone call, particularly via an assessment of the modified Rankin score.

SUMMARY:
Study like register with biomarkers samples for patient experiencing acute ischemic stroke, to assess clinical outcomes and different factors that may affect the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older (i.e., candidates must have had their 18th birthday)
* Neuroimaging demonstrates acute ischemic stroke with large vessel proximal with the use of neuro-thrombectomy devices intended to restore blood flow
* No upper or lower limits of the neurological severity at baseline (NIHSS).
* With or without intravenous thrombolysis
* Oral informed consent (patient and/or trustworthy person)

Non-inclusion Criteria:

* Pregnant or breast-feeding women
* Patient benefiting from a legal protection
* Non-membership of a national insurance scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with stroke treated by thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | Day 90
  modified Rankin score (mRS), score 0 to 6 with 0 = no symptoms and 6 = death.

SECONDARY OUTCOMES:
Efficacy on reperfusion (modified Thrombolysis in Cerebral Infarction (mTICI) 2b/3) | Day 1
  Rate of complete or near complete reperfusion (modified Thrombolysis in Cerebral Infarction (mTICI) 2b/3)
Efficacy on revascularization (>= mTICI 2b) | Day 1
  Time to achieve TICI 2b or better revascularization
Efficacy on clinical outcome (mRS=0-1) | Day 90
  Rate of excellent functional outcome defined as a modified Rankin score (mRS) 0-1
Efficacy on functional independence (mRS 0-2) | Day 90
  Rate of functional independence defined as a modified Rankin score 0-2
Hemorrhage evaluated by imagery | Day 0
  Rate of symptomatic and asymptomatic intracerebral hemorrhage at MRI or CT scan
Hematoma rate | Day 1
  Rate of parenchymal hematoma 2
Mortality rate | Day 90
  Rate of all-cause mortality
Complication rate | Day 0
  Rate of periprocedural complications
ASPECT (Alberta Stroke Program Early CT score) | Day O
  Measure by Axial imaging, 10-point quantitative topographic CT scan score
Parametric imaging | Day 0
  Diffusion, volume clinical-diffusion mismatch
Imaging data | Day 1
  Angiographic imaging
Blood sampling for research purpose | Day 0
  Search of biomarkers of stroke etiology and recovery

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Larpergue, MD, Principal Investigator — Hopital Foch
Locations (16):
- France (16):
  - CHU Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - Hôpital le Kremlin-Bicètre - APHP, Le Kremlin-Bicêtre
  - CHU Dupuytren, Limoges
  - CHU Lyon, Lyon
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hôpital Pitié Salpétrière, Paris
  - Hôpital SAINTE ANNE, Paris
  - Fondation Ophtalmique de Rotschild, Paris
  - CHU Rennes, Rennes
  - Chu Rouen, Rouen
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milnerowicz M, Desilles JP, Pop R, Dargazanli C, Labreuche J, Sibon I, Gory B, Soize S, Bourcier R, Mazighi M, Cognard C, Caroff J, Gentric JC, Clarencon F, Richter S, Janot K, Lapergue B, Marnat G; ETIS investigators. Cangrelor versus GPIIb/IIIa inhibitors as adjunctive therapy in endovascular treatment of large vessel occlusion stroke. J Neurointerv Surg. 2025 May 2:jnis-2025-023260. doi: 10.1136/jnis-2025-023260. Online ahead of print. PMID 40316319
- [Derived] Dargazanli C, Mourand I, Mahmoudi M, Poirier L, Labreuche J, Weisenburger-Lile D, Gory B, Richard S, Ducroux C, Piotin M, Blanc R, Lucas L, Marnat G, Aubertin M, Arquizan C, Bourcier R, Detraz L, Vannier S, Guillen M, Eugene F, Walker G, Lun R, Dowlatshahi D, Shamy M, Consoli A, Costalat V, Lapergue B, Maier B, Guenego A, Fahed R. Endovascular treatment versus medical management for basilar artery occlusion with low-to-moderate symptoms (National Institutes of Health Stroke Scale < 10). Eur Stroke J. 2025 Jun;10(2):397-405. doi: 10.1177/23969873241290442. Epub 2024 Oct 13. PMID 39397363
- [Derived] Derraz I, Moulin S, Gory B, Kyheng M, Arquizan C, Costalat V, Lapergue B; ETIS Investigators. Endovascular Thrombectomy Outcomes with and without Intravenous Thrombolysis for Large Ischemic Cores Identified with CT or MRI. Radiology. 2023 Oct;309(1):e230440. doi: 10.1148/radiol.230440. PMID 37847131
- [Derived] Malka D, Janot K, Pasi M, Desilles JP, Marnat G, Sibon I, Consoli A, Dargazanli C, Arquizan C, Gory B, Richard S, Naggara O, Clarencon F, Rosso C, Bourcier R, Eker O, Caroff J, Lapergue B, Boulouis G; ETIS collaborators. Effects of weather conditions on endovascular treatment case volume for patients with ischemic stroke. J Neuroradiol. 2023 Nov;50(6):593-599. doi: 10.1016/j.neurad.2023.07.001. Epub 2023 Jul 11. PMID 37442271
- [Derived] Bourcier R, Consoli A, Desilles JP, Labreuche J, Kyheng M, Desal H, Alias Q, Gory B, Dargazanli C, Janot K, Zhu F, Lapergue B, Marnat G. Temporal trends in results of endovascular treatment of anterior intracranial large cerebral vessel occlusion: A 7-year study. Eur Stroke J. 2023 Sep;8(3):655-666. doi: 10.1177/23969873231180338. Epub 2023 Jun 8. PMID 37288701
- [Derived] Douarinou M, Gory B, Consoli A, Lapergue B, Kyheng M, Labreuche J, Anadani M, Blanc R, Marnat G, Bourcier R, Sibon I, Eugene F, Vannier S, Audibert G, Mione G, Richard S; ETIS Investigators. Impact of Strategy on Clinical Outcome in Large Vessel Occlusion Stroke Successfully Reperfused: ETIS Registry Results. Stroke. 2022 Jan;53(1):e1-e4. doi: 10.1161/STROKEAHA.121.034422. Epub 2021 Nov 3. PMID 34727741
- [Derived] Happi Ngankou E, Gory B, Marnat G, Richard S, Bourcier R, Sibon I, Dargazanli C, Arquizan C, Maier B, Blanc R, Lapergue B, Consoli A, Vannier S, Spelle L, Denier C, Boulanger M, Gauberti M, Saleme S, Macian F, Clarencon F, Rosso C, Naggara O, Turc G, Ozkul-Wermester O, Papagiannaki C, Viguier A, Cognard C, Lebras A, Evain S, Wolff V, Pop R, Timsit S, Gentric JC, Bourdain F, Veunac L, Eugene F, Finitsis S; ETIS Registry Investigatorsdagger. Thrombectomy Complications in Large Vessel Occlusions: Incidence, Predictors, and Clinical Impact in the ETIS Registry. Stroke. 2021 Dec;52(12):e764-e768. doi: 10.1161/STROKEAHA.121.034865. Epub 2021 Oct 28. PMID 34706564
- [Derived] Aubertin M, Weisenburger-Lile D, Gory B, Richard S, Blanc R, Ducroux C, Piotin M, Labreuche J, Lucas L, Dargazanli C, Benali A, Bourcier R, Detraz L, Vannier S, Guillen M, Eugene F, Walker G, Lun R, Guenego A, Consoli A, Marnat G, Maier B, Lapergue B, Fahed R; ETIS Investigators*. First-Pass Effect in Basilar Artery Occlusions: Insights From the Endovascular Treatment of Ischemic Stroke Registry. Stroke. 2021 Dec;52(12):3777-3785. doi: 10.1161/STROKEAHA.120.030237. Epub 2021 Aug 26. PMID 34433309
- [Derived] Ducroux C, Renaud N, Bourcier R, Marnat G, Sibon I, Gory B, Richard S, Dargazanli C, Arquizan C, Eugene F, Vannier S, Labreuche J, Walker G, Blanc R, Obadia M, Consoli A, Lapergue B, Fahed R; ETIS investigators. Embolus Retriever with Interlinked Cages (ERIC) versus conventional stent retrievers for thrombectomy: a propensity score-based analysis. J Neurointerv Surg. 2021 Mar;13(3):255-260. doi: 10.1136/neurintsurg-2020-016289. Epub 2020 Jun 30. PMID 32606101
- [Derived] Boisseau W, Fahed R, Lapergue B, Desilles JP, Zuber K, Khoury N, Garcia J, Maier B, Redjem H, Ciccio G, Smajda S, Escalard S, Taylor G, Mazighi M, Michel P, Gory B, Blanc R; ETIS Investigators. Predictors of Parenchymal Hematoma After Mechanical Thrombectomy: A Multicenter Study. Stroke. 2019 Sep;50(9):2364-2370. doi: 10.1161/STROKEAHA.118.024512. Epub 2019 Jul 22. PMID 31670928